

# DEPARTMENT OF INTERNAL MEDICINE UNIVERSITI KEBANGSAAN MALAYSIA

Official Title: A Randomised, Open Label, Interventional Study Evaluating the Efficacy & Safety of Dry Powder Ivy Extract (Syrup Prospan) versus NAC among COPD Patients

### (SyProNAC Trial)

Research Identification Number: FF-2023-433 Date of Document: Version 1st February 2024

### Candidate:

Dr Muhamad Thaqif Sidek

(P126274)

### **Supervisor:**

Dr Mas Fazlin Mohamad Jailaini
Respiratory Unit, Department of Medicine, HCTM

### **Co-supervisor:**

Associate Professor Dr Mohamed Faisal Abdul Hamid Associate Professor Dr Andrea Ban Yu-Lin Dr Azat Azrai Dato Azmel Dr Ng Boon Hau Dr Nik Nuratiqah Nik Abeed Respiratory Unit, Department of Medicine, HCTM

| CONTENTS | PAGE |
|---|---|
| Section 1: Introduction | 3 |
| Section 2: Literature Review | 4 |
| Section 3: Hypothesis | 6 |
| Section 4: Research Objectives | 6 |
| Section 5: Research design & methodology 5.1 Study Design 5.2 Study Population 5.3 Inclusion and Exclusion Criteria 5.4 Study Protocol and Data Acquisitions 5.5 Operational Terms Definition 5.6 Sample Size and Power of Study | 7 |
| Section 6: Statistical Analysis | 13 |
| Section 7: Research Ethics | 14 |
| Section 8: Estimated Cost of Study | 15 |
| Section 9: Research Information | 16 |
| Section 10: Consent Form | 20 |
| Section 11: Data Collection Sheet | 22 |
| Section 12: Gantt chart | 24 |
| Section 13: Appendices | 25 |
| Section 14: References | 30 |

#### **Section 1: Introduction**

As the third global leading cause of death, Chronic Obstructive Pulmonary Disease (COPD) affects more than 300 million people worldwide [1,2]. These patients suffer from 0.5–3.5 exacerbations per year on average. Each exacerbations dampened their health status as well as quality of life, not to mention a great burden to our healthcare system [3,4]. Those partially treated or prolonged exacerbations would subsequently lead to unfavorable disease progression. Hence a holistic approach in managing each exacerbations is very crucial [5].

Mucus hypersecretion in COPD patients plays a pivotal role in acute exacerbations and associated with unfavorable outcomes [6]. These exacerbations comes with sputum increment as much as its purulence. Mucolytics are believed to to ease patient to expectorate and benefits them from tip into an exacerbations or even the consequent hospitalisation [7].

Mucolytics work by reducing sputum viscosity hence improved its expectoration. N-acetylcysteine (NAC) is a mucolytic with antioxidant and anti-inflammatory properties, commonly used in practice among COPD patients [8]. Meanwhile, Syrup Prospan is ivy leaf preparations, obtained as extracts from leaves of the plant Hedera helix L. It is widely used over-the-counter cough remedy containing saponins which are believed to have expectorant properties [9]. Studies show evidence of antispasmodic, bonchodilating, anti-inflammatory and antitussive properties and its usage is authorised by the European Medicines Agency [10].

#### **Section 2: Literature Review**

Mucolytics are defined as medications that decrease mucus viscosity and can be divided into classic and peptide mucolytics. Classic and peptide mucolytics depolymerize mucin glycoproteins and DNA with F-actin polymer networks, respectively [11].

NAC alters mucus viscosity by modifying the crosslinks and molecular interactions within mucin polymers. These changes enhancing mucociliary clearance and subsequent sputum expectoration. This effects are beneficial in mucus hypersecretory states such as COPD and cystic fibrosis.

Several studies on NAC suggest apart from its mucolytic properties, it exerts anti-inflammatory effects by inhibiting chemotaxis, reducing lysozymes and lactoferrin concentration as well as neutrophils and macrophages in bronchoalveolar lavage fluid [12]. In addition, it inhibits bacterial adherence to the ciliated epithelium [13].

Latest 2023 GOLD Report stated that COPD patients not receiving ICS, regular treatment with mucolytics such as carbocysteine and N-acetylcysteine (NAC) may reduce exacerbations and modestly improve health status.

A meta-analysis by Papadopoulou et al included 24 RCTs involving 2192 patients with COPD exacerbations demonstrated with moderate certainty that mucolytics appear to improve the treatment success rate and symptoms [14].

Another meta analysis conducted by Cazzola et al demonstrates that mucolytics are useful in preventing COPD exacerbations as maintenance add-on therapy to patients with frequent exacerbations. The effectiveness of mucolytics is independent of the severity of airway obstruction and the use of inhaled corticosteroids [15].

Various trials proved the efficacy and safety of ivy leaves preparation for acute URTI and also chronic bronchitis. Schaefer et al proved consistent superiority of ivy leaves cough liquid in a randomized, placebo-controlled, double-blind trial [16]. A cohort study in Germany provided further evidence that the use of ivy leaves preparations contribute to inappropriate antibiotic usage for respiratory infections in adult patients with cough symptoms [17].

To date there are no studies comparing Ivy leaf preparations with other mucolytic agents. A meta analysis by Rogliani et al assessed the efficacy of erdosteine, carbocysteine, and NAC on acute exacerbation and concluded that overall efficacy and safety profile of erdosteine is superior to that of both carbocysteine and NAC [18].

### **Section 3: Hypothesis**

- 1. Syrup Prospan is non inferior to NAC no significant difference of cough symptoms and its impact on daily activities, health related quality of life, as well as lung function test at 30 days of treatment
- 2. Patients received Syrup Prospan has higher satisfaction score compared to N-Acetylcysteine

### **Section 4: Research Objectives**

### **Primary objective**

To demonstrate that Syrup Prospan is non inferior to N-Acetylcysteine in assessment of cough symptoms and its impact on daily activities using Cough and Sputum Assessment Questionnaire (CASA-Q) during 30 days of treatment.

### **Secondary objective**

- 1. To evaluate the effectiveness of Syrup Prospan vs N.Acetylcysteine in terms of
  - I. McGill COPD Quality of Life Questionnaire on Day 1 and 30 days of treatment.
  - II. Lung function test (including morning pre-dose FEV1) and FVC on Day 1 and 30 days of treatment.
  - III. Incidence of adverse effects (in %)
- 2. To assess satisfaction of treatment using the 5 point Likert Scale.

### **Section 5: Research Design & Methodology**

### 5.1 Study Design

A randomised, open label, interventional study evaluating the efficacy and safety of dry powder Ivy Extract (Syrup Prospan) versus NAC among COPD patients.

Randomization 1:1 to received either N.Acetylcysteine 600 mg BD or Syrup Prospan 7.5mls BD (Block randomization)

### 5.1.1 Period of Study

The study will be conducted from December 2023 to November 2026 after receiving approval by the research ethics committee.

### 5.2 Sampling Population

This study will include All patients are stable COPD patients under Respiratory Clinic HCTM follow-up, aged  $\geq$  40 year old and above and able to perform spirometry from September 2023 to February 2024. Demographic and clinical data will be collected. Patient will be followed-up at Day 15 and Day 30 after intervention.

#### 5.3 Inclusion and Exclusion Criteria

#### **Inclusion criteria**

- 1. Patients with documented post bronchodilator FEV1/FVC < 70 or <LLN
- 2. Age 40 years and above
- 3. Able to perform spirometry
- 4. Patient with Stable COPD based on GOLD 2023 strategy

#### **Exclusion criteria**

- 1. Diagnosis of other chronic lung diseases: Asthma, Asthma-COPD Overlap, Interstitial Lung Disease, Bronchiectasis, Lung Cancer
- 2. Patients with contraindication for spirometry: recent cardiac complications, major surgery, severe advanced respiratory disease, or those with cognitively or neurologically impairment
- 3. Hypersensitivity to acetylcysteine or any component of the formulation
- 4. Hypersensitivity to dry powder ivy extract
- 5. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG (human Chorionic Gonadotropin) laboratory test
- 6. Patients on pre-existing regular mucolytics (at least 1 month prior)
- 7. Illiterate patients

### 5.4 Study Protocol and Data Acquisitions

This is a prospective interventional study conducted on COPD patients under the Respiratory Unit, Department of Internal Medicine in HCTM, who qualified both the inclusion and exclusion criteria. Patients will be briefed about this study.

Subsequently, consent will be obtained from those who are agree to participate from the patient him/herself.

Patients' will be assessed first with several modalities particularly spirometry, CAT score, McGill COPD Quality of Life and Cough and Sputum Assessment Questionnaire (CASA-Q) prior to the commencement of treatment. Patients will be seen on Day 15 to evaluate patients' adherence, compliance as well as adverse effect. Then patients will be assessed again on Day 30 of treatment with the same set of evaluation tools as in the beginning of the study.

### 5.4.1 Recruitment/Data Collection Pathway



### 5.5 Operational Term Definitions

### Stable COPD based on GOLD 2023 strategy

All outpatient COPD patients, GOLD I, II, III, IV as per GOLD 2023 Guidelines seen in Respiratory Clinic HCTM and not in exacerbation upon recruitment

### **Exacerbation (as per GOLD Executive Summary)**

An event in the natural course of the disease characterise by change in the patient's baseline dyspnoea, cough and/or sputum beyond normal day-to-day variation that is acute onset and may warrant change in regular medications

### Adherence and compliance

Using pill count method, the adherence rate is determined by the following formula

% adherence = (Quantity dispensed) - (Quantity remaining) / (Prescribed no of tablets/day) x (No of days between dispensing date and interview)

For Syrup Prospan we will quantify by determine the volume of syrup

#### **Adverse Effects**

Any desirable effects that experienced by patients after started on the aforementioned medication

### 5.6 Sample Size and Power of Study

In order to calculate the required sample size, we will employ the Cohen's d formula for estimating the effect size (Cohen, 1988) [19]. The formula is given as

$$d = \frac{M_1 - M_2}{\sqrt[2]{\frac{SD_1^2 + SD_2^2}{2}}}$$

Where d is the Cohen's effect size, M<sub>1</sub> and M<sub>2</sub> are the mean for the first and second group, and SD<sub>1</sub> and SD<sub>2</sub> are the standard deviation for the first and second group respectively. Based on a similar study by Kuzmenko et al. (2020) [20] which employs the CAT score to assess the efficacy of NAC in patients with COPD, the mean and standard deviation for before and after treatment are given as:

Before treatment:  $23.46 \pm 3.66$ After treatment:  $20.38 \pm 5.78$ 

Hence, this give the values of  $M_1 = 23.46$  and  $M_2 = 20.38$ , and  $SD_1 = 3.66$  and  $SD_2 = 5.78$  that can use to estimate the effect size using the formula above.

$$d = \frac{23.46 - 20.38}{\sqrt[2]{\frac{3.66^2 + 5.78^2}{2}}} = 0.637$$

Therefore, it gives an estimated effect size of 0.637 which is considered to be a medium effect size.

With a power of 80% and a level of significance of 5% for detecting an effect size of 0.637, we calculate the required

sample size using an online sample size calculator (Dhand & Khatkar, 2014) [21] for comparing paired differences. It gives at a value of 23 participants for each group which mean the required number of participants is 46.

Additional of 20% samples is recruited to avoid missing data due to withdrawal or drop out. Therefore, a total of minimum 55 patients will be recruited for this study. However, we aim to recruit 100 patients for our study where the treatment is given to equal number of participants in each group.

### **Section 6: Statistical Analysis**

Data were collected manually with a data collection sheet. Demographic data and patient characteristic will be analysed using descriptive analysis and Chi-square method. Continuous variables were presented as mean  $\pm$  SD and categorical variables as percentages, unless stated otherwise.

All statistical analysis for the study will be performed using statistic software SPSS version 24.0 (IBMSPSS Statistics 2017). A p-value of <0.05 is considered statistically significant.

#### **Section 7: Research Ethics**

Approval from the Research and Ethics Committee of Hospital Canselor Tuanku Muhriz onbtained with research code FF-2023-433. All the collected information will be strictly confidential and only accessible by the research team members. All patients will be kept anonymous and coded into the data collection sheet.

Participant will only be recruited in this study if informed consent was given, and will be allowed to withdraw from the study at any point. The research will be conducted according to standard of good clinical practice and the rights and safety of the participants are guaranteed throughout the study.

## **Section 8: Estimated Cost of Study**

| ACTIVITY /<br>DEVICE | AMOUNT | COST<br>PER<br>ITEM | ESTIMATED COST |
|---|---|---|---|
| Syr Prospan 7.5ml | 450ml (4 and | RM18.9 | RM4725 |
| BD | half bottle) x | per | |
| (Sponsored by | 50 patients | bottle | |
| DELFI) Tab NAC 600mg | 60 tablets x 50 | RM3.29 | RM9870 |
| BD | patients | per | 14,15,07,0 |
| (Sponsored by | | tablet | |
| DELFI) | | | |
| Printing: | | | |
| i) Research | 2 pages for | RM0.40 | RM48 |
| Information | each set x 100 | | |
| ii) Consent form | 1 page for | RM0.20 | RM24 |
| | each set x 100 | KIVIU.20 | KW124 |
| iii) Data | | | |
| collection | 2 pages for | RM0.40 | RM48 |
| sheet | each set x 100 | | |
| Silect | caen set a 100 | | |
| iv) CAT Score | 1 page for | | |
| Questionnaire | each set x 100 | RM0.20 | RM24 |
| Questionnaire | cacii set x 100 | | |
| v) McGill COPD | 6 pages for | RM1.20 | RM144 |
| QoL | each set x 100 | 10.11.20 | |
| Questionnaire | Cucii bet A 100 | | |
| Questionnane | | | |
| TOTAL ES | <br>TIMATED COS | <u> </u><br>T | RM14883 |

#### **Section 9: Research Information Sheet**



#### Research Title:

A Randomised, Open Label, Interventional Study Evaluating the Efficacy & Safety of Dry Powder Ivy Extract (Syrup Prospan) versus NAC among COPD Patients

#### Researcher's Name:

Dr Mas Fazlin Mohamad Jailaini / Dr Muhamad Thaqif bin Sidek

#### Place of Conduct:

Respiratory Unit, Department of Internal Medicine, Hospital Canselor Tuanku Muhriz

#### Introduction:

COPD is a progressive airway disease and mucolytics help controlling symptoms as well as prevent future exacerbations.NAC is a common mucolytic agent and Syrup Prospan is ivy leaf preparations used to serve this purpose.

#### Purpose of Study:

This study aims to evaluating the efficacy and safety of Ivy Extract preparations against NAC as mucolytic in COPD patients.

#### Type of Intervention:

You will be randomised either in 'Interventional group' or 'non-interventional group'. For the interventional group, we will change your mucolytic agent to Syrup Prospan. For the non-interventional group, we will continue your current NAC. We will first get a baseline spirometry, CAT score, McGill COPD QoL Questionnaire and CASA-Q on D1. We will continue follow-up closely for both group and assess your adherence to medications and adverse effects on D15 and finally on D30 of treatment with repeat spirometry, CAT score, McGill COPD QoL Questionnaire and CASA-Q.

Risk of joining in this study:

- There are no surgical intervention / life threatening side effects involved with this study, therefore no major risk is associated upon enlistment.
- The documented side effects for both medications are as follows;
  - o NAC anaphylaxis; skin rash, urticaria, bronchospasm, angioedema
  - o Ivy Leaf Extract nausea, vomiting, diarrhoea, allergic reaction

<sup>\*</sup>If you experiences any side effects other than mentioned above, kindly inform us for subsequent appropriate measures.

Participation in this study is entirely voluntary. It is your choice to participate (or allow patient to participate). Regardless of your choice, the standard quality of care and treatment remain the same. All data obtained will be recorded and will be used for analysis.

#### **Confidentiality:**

Information collected during this study will be kept confidential. Access to the data is only by the researcher team and the Research Ethics Committee of HCTM. No specific reference to any individual will be reported in this study. Participants have the right to know the outcome of this study.

#### Reimbursements:

Participants do not have to pay for the spirometry, nor be paid for participating in this study.

#### Right to Refuse or Withdraw:

This study is of voluntary basis, patient or his/her next-of-kin have the right to withdraw from this study at any time of the study. The choice is yours and all your right will be respected.

### **Section 10: Consent Form**

| R | esear | ·ch | Tif | le |
|---|-------|-----|-----|----|

DATE:

A Randomised, Open Label, Interventional Study Evaluating the Efficacy & Safety of Dry Powder Ivy Extract (Syrup Prospan) versus NAC among COPD Patients

| R | esea | rch | er's | No | me | ٠. |
|---|------|-----|------|----|----|----|

| Researcher's Name: |
|---|
| Dr Mas Fazlin Mohamad Jailaini / Dr Muhamad Thaqif bin Sidek |
| I,, |
| IC No:, |
| <ul> <li>Have read all the information in the Patient Information Sheet and understand the aim and purpose of this study.</li> <li>Have been given enough time to think about it and all of my question have been answered to my satisfaction.</li> <li>Understand that I may freely choose to withdraw from this study at any time without reason and without repercussions.</li> <li>Understand that anonymity will be ensured in the final write up.</li> <li>I understand all the above and voluntarily agree to take part in this research study, to follow the study procedures and to provide the necessary information as requested.</li> </ul> |
| Signature/Thumbprint DATE: |
| Witness Name/IC no:<br>DATE: |

Researcher Name/IC no: Dr Muhamad Thaqif Sidek (900617-10-6037)

## **Section 11: Data Collection Sheet**

Patient's Sticker

| Contact Number: | •••••• |
|-----------------------------|--------|
| Age: | •••••• |
| Gender: | •••••• |
| Ethnicity: | ••••• |
| Background Medical Problem: | |
| Diabetes Mellitus | |
| • Hypertension | |
| • Ischaemic heart Disease | |
| • Heart Failure | |
| • Previous stroke | |
| • Dyslipidaemia | |
| • Others: | •••••• |
| Weight: | |
| Height: | |
| BMI: | |
| First diagnosis of COPD: | |
| MMRC: | ••••• |
| . A . SCHIP. | |

| year: | ns in the past 1 | ••••• |
|---|---|---|
| Date of recent spiromet | try: | ••••• |
| FEV1 (post-bronchodil | ator): | ••••• |
| Types of inhalers: | | |
| Inhaler technique: Correct | Incorrect | |
| | D1 | D30 |
| Spirometry | | |
| CAT score | | |
| McGill COPD QoL | | |
| CASA-Q | | |
| Adherence: | ••••••••••••••••••••••••••••••••••••••• | ••••••••••••••••••••••••••••••••••••••• |
| Adverse effects: | ••••• | ••••• |

### **Section 12: Gantt Chart**

| Progression / Timeline | Mac<br>2023 -<br>May<br>2023 | Jun<br>2023 -<br>Oct<br>2023 | Dec 2023 | Jan<br>2024<br>- Dec<br>2024 | Dec<br>2024<br>- Dec<br>2025 | Jan<br>2026<br>- Oct<br>2026 | Nov<br>2026 |
|---|---|---|---|---|---|---|---|
| Literature review | | | | | | | |
| Proposal preparation,<br>correction and<br>presentation to Medical<br>Department, UKMMC | | | | | | | |
| Approval of UKMMC<br>Research and Ethics<br>Committee | | | | | | | |
| Patient recruitment | | | | | | | |
| Data entry and analysis | | | | | | | |
| Final result and manuscript submission | | | | | | | |
| Thesis presentation | | | | | | | |

## **Section 13: Appendices**

| Your name: | | Today's date: COPD Assessment Test |
|---|---|---|
| How is your COP | D? Take the COPD A | ssessment Test™ (CAT) |
| Pulmonary Disease) is having on | your well being and daily life. Your answe | re the impact COPD (Chronic Obstructive<br>ers, and test score, can be used by you and<br>D and get the greatest benefit from treatment. |
| For each item below, place a mark<br>for each question. | | urrently. Be sure to only select one response |
| Example: I am very happy | 0 🔏 2 3 4 5 | I am very sad SCORE |
| I never cough | 012345 | I cough all the time |
| I have no phiegm (mucus)<br>in my chest at all | 012345 | My chest is completely full of phlegm (mucus) |
| My chest does not<br>feel tight at all | 012345 | My chest feels very tight |
| When I walk up a hill or<br>one flight of stairs I am<br>not breathless | 012345 | When I walk up a hill or one flight of stairs I am very breathless |
| I am not limited doing any activities at home | 012345 | I am very limited doing activities at home |
| I am confident leaving<br>my home despite my<br>lung condition | 012345 | I am not at all confident<br>leaving my home because<br>ofmy lung condition |
| I sleep soundly | 012345 | I don't sleep soundly<br>because of my lung<br>condition |
| I have lots of energy | 012345 | I have no energy at all |
| COPD Assessment Test and the CAT lo<br>© 2009 GlaxoSmithKine group of compo<br>Last Updated: February 24, 2012 | go is a trade mark of the GlaxioSmithKline group o<br>anies. All rights reserved. | companies. TOTAL SCORE |

| | | McGill COPD Quality of Life Questionnaire | |
|---|---|---|---|
| Cent | re L | Project Visit Visit | |
| Pre-r | ehabilitation ev | valuation (visit 1) Post-rehabilitation evaluation < 1 month (visit 2) | |
| Post- | rehabilitation e | evaluation : 1 yr (visit 3) 2 yrs (visit 4) 3 yrs (visit 5) | |
| Date | | yyyy-mmm-dd Time at the beginning of the questionnaire | on 24:00 |
| | | tly has or had an exacerbation in the past 4 weeks? No Yes | |
| | nptoms | | |
| | iptoms<br>How much fa | atique have you experienced in the last four weeks? | |
| | ptoms How much fa | latique have you experienced in <u>the last four weeks</u> ? No fatigue at all Some fatigue | |
| | How much fa | latique have you experienced in the last four weeks? No fatigue at all Some fatigue Moderate fatigue | |
| | uptoms How much fa 1- 2- 3- 4- | Tatique have you experienced in the last four weeks? No fatigue at all Some fatigue Moderate fatigue A lot of fatigue | |
| 1- | How much fa<br>1-<br>2-<br>3-<br>4-<br>5- | latique have you experienced in the last four weeks? No fatigue at all Some fatigue Moderate fatigue | |
| 1- | How much fa<br>2-<br>3-<br>4-<br>5-<br>On an averag | Tatique have you experienced in the last four weeks? No fatigue at all Some fatigue Moderate fatigue A lot of fatigue Extreme fatigue | |
| 1- | How much fa<br>1-<br>2-<br>3-<br>4-<br>5-<br>On an averag | Tatique have you experienced in the last four weeks? No fatigue at all Some fatigue Moderate fatigue A lot of fatigue Extreme fatigue | |
| 1- | How much fa<br>1-<br>2-<br>3-<br>4-<br>5-<br>On an averag | Tatique have you experienced in the last four weeks? No fatigue at all Some fatigue Moderate fatigue A lot of fatigue Extreme fatigue ge day during the past four weeks, Nerver | |
| 1- | How much fa 1- 2- 3- 4- 5- On an average 1- 2- 3- 4- | Valique have you experienced in the last four weeks? No fatigue at all Some fatigue Moderate fatigue A lot of fatigue Extreme fatigue ge day during the past four weeks, Nerver A few times Some times Many times | |
| 1- | How much fa 1- 2- 3- 4- 5- On an average 1- 2- 3- 4- | No fatigue at all Some fatigue Moderate fatigue A lot of fatigue Extreme fatigue Age day during the past four weeks, Nerver A few times Some times | |
| 1- | How much fa 1- 2- 3- 4- 5- On an averag | Valique have you experienced in the last four weeks? No fatigue at all Some fatigue Moderate fatigue A lot of fatigue Extreme fatigue ge day during the past four weeks, Nerver A few times Some times Many times | |

| | <ul><li>No shortness of breath</li><li>Very little shortness of breath</li></ul> | | | | | |
|---|---|---|---|---|---|---|
| | 3- Moderate shortness of breath | | | | | |
| | 4- A lot of shortness of breath | | | | | |
| | 5- Extreme shortness of breath | | | | | |
| | a. Doing you normal daily activities. | | | | | |
| | b. Performed activities that required you to raise | your arms o | verhead. | | | |
| | c. Walking on the level at your own pace. | | | | | |
| _ | | | | | | |
| e | eling A | | | | | |
| - | During the <u>last four weeks</u> , how often <u>did the</u> activities of daily life? | fear of becor | ming short o | f breath limi | t you in yo | ur |
| | 1- All of the time | | | | | |
| | 2- Many times | | | | | |
| | 3- Some of the times | | | | | |
| | 4- A few times | | | | | |
| | 4- A few times | | | | | |
| | 4- A few times<br>5- None of the time | often have j | you felt: | | | |
| | 4- A few times<br>5- None of the time | often have | you felt: | | | |
| <b>i-</b> | 4- A few times<br>5- None of the time | often have | you felt: | Some of | A few | None of |
| i- | A few times None of the time On an average day in the past four weeks how | | | Some of<br>the times | A few times | None of the time |
| - | A few times None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to | All of the | Many of | | | |
| - | A few times None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. | All of the time | Many of<br>the times | the times | times<br>4 | the time |
| j- | A few times None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to | All of the time | Many of the times | the times | times | the time |
| - | A few times None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. | All of the time | Many of<br>the times | the times | times<br>4 | the time |
| 1- | A few times None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. | All of the time | Many of the times | the times 3 | times<br>4 | the time |
| 5- | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. | All of the time | Many of the times | 3 3 3 | times 4 4 4 | the time 5 5 5 |
| | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. Unable to accept your pulmonary condition. | All of the time | Many of the times | 3 3 3 | times 4 4 4 | the time 5 5 5 |
| el | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. Unable to accept your pulmonary condition. | All of the time 1 1 1 1 | Many of the times 2 2 2 2 | 3 3 3 3 | 4 4 4 4 | 5 5 5 5 |
| eli | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. Unable to accept your pulmonary condition. | All of the time 1 1 1 1 w things have | Many of the times 2 2 2 2 ve been with | 3 3 3 3 you during a | times 4 4 4 4 the past 4 | 5 5 5 5 weeks. |
| el | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. Unable to accept your pulmonary condition. | All of the time 1 1 1 w things have that comes of | Many of the times 2 2 2 2 ve been with | 3 3 3 3 you during a | times 4 4 4 4 the past 4 | 5 5 5 5 weeks. |
| el | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. Unable to accept your pulmonary condition. Iling B These questions are about how you feel and hor for each question, please give the one answer. | All of the time 1 1 1 1 w things have that comes | Many of the times 2 2 2 2 2 Most of the times | 3 3 3 3 you during a way you ha | 4 4 4 4 the past 4 tive been fe | the time 5 5 5 5 weeks. |
| el | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. Unable to accept your pulmonary condition. Iling B These questions are about how you feel and hor for each question, please give the one answer. | All of the time 1 1 1 1 w things have that comes of | Many of the times 2 2 2 2 2 ve been with losest to the | 3 3 3 3 you during a way you ha | 4 4 4 4 4 A the past 4 ve been fe | the time 5 5 5 5 None of the |
| el | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. Unable to accept your pulmonary condition. Iling B These questions are about how you feel and hor for each question, please give the one answer. | All of the time 1 1 1 1 w things have that comes | Many of the times 2 2 2 2 2 Most of the times | 3 3 3 3 you during a way you ha | 4 4 4 4 the past 4 tive been fe | the time 5 5 5 5 weeks. |
| el | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. Unable to accept your pulmonary condition. Iling B These questions are about how you feel and hor for each question, please give the one answer. | All of the time 1 1 1 1 w things have that comes | Many of the times 2 2 2 2 2 Most of the times | 3 3 3 3 you during a way you ha | 4 4 4 4 4 A the past 4 ve been fe | the time 5 5 5 5 None of the |
| el | 4- A few times 5- None of the time On an average day in the past four weeks how Fringhtened or worried about not being able to breathe. Frustrated or impatient. That everything seems too much of an effort. Unable to accept your pulmonary condition. ling B These questions are about how you feel and hor for each question, please give the one answer thow much of the time during the past 4 weeks. | All of the time 1 1 1 1 1 All the time | Many of the times 2 2 2 2 2 Most of the time | 3 3 3 3 you during a way you ha | times 4 4 4 4 4 the past 4 ve been fe A little of the time | the time 5 5 5 5 None of the time |

| c. | Have you felt downhearted and depressed? | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|---|
| d. | Did you feel worn out? | 1 | 2 | 3 | 4 | 5 |
| <b>7</b> | How TRUE or FALSE is each of the following My health is excellent. | Definitely true | Mostly true | Don't<br>know | Mostly<br>false | Definite<br>ly false |
| Ph | ysical Function A | | | | | |
| 8 | daily activities? 1- Not at all longer 2- Somewhat longer 3- Moderately longer 4- Quite a bit longer | much more time | does it ta | ke <u>you to per</u> | <u>form your</u> | |
| 9 | daily activities ? 1- Not at all longer 2- Somewhat longer 3- Moderately longer 4- Quite a bit longer 5- A lot longer | u might do <u>durir</u><br>ability to perform<br>Not limited | ng a typica<br>n these act | <u>l day</u> . To who<br>ivities ?<br>Moderately | at extend d | Extremel |
| 9 | daily activities ? 1- Not at all longer 2- Somewhat longer 3- Moderately longer 4- Quite a bit longer 5- A lot longer | u might do <u>durir</u><br>ubility to perforn | ng a typica<br>n these act | <u>l day</u> . To wha<br>ivities ? | nt extend d | - |
| | daily activities? 1. Not at all longer 2. Somewhat longer 3. Moderately longer 4. Quite a bit longer 5. A lot longer The following items are about activities yo breathing problems now limit you in your a | u might do <u>durir</u><br>bblity to perform<br>Not limited<br>at all | n <u>g a typica</u><br>n these act<br>Limited<br>a little | <u>l daγ</u> . Το wha<br>iivities ?<br>Moderately<br>limited | at extend d | Extremel<br>limited |

#### Physical Function B

Being autonomous in your own home ie. not requiring any assistance.

Being able to function sexually (If sexual activity is not an issue for you, answer « not limited at all »)

10 The following items are about activities you might do <u>during a typical day</u>. Does your <u>health now limit you</u> in these activities? If so, how much?

2

3

3

| | | Not limited at all | Limited a little | Moderately<br>limited | Limited a lot | Extremel |
|---|---|---|---|---|---|---|
| a. | Climbing one flight of stairs. | 1 | 2 | 3 | 4 | 5 |
| b. | Bending, kneeling, or stooping. | 1 | 2 | 3 | 4 | 5 |
| C. | Walking more than a kilometer. | 1 | 2 | 3 | 4 | 5 |
| | work or other daily activities as a result of | All the time | Most of the time | Some of the time | A little of the time | None of the time |
| a. | Cut down the <b>amount of time</b> you spent on work or other activities | 1 | 2 | 3 | 4 | 5 |
| b. | Accomplished less than you would like | 1 | 2 | 3 | 4 | 5 |
| C. | Had <b>difficulty</b> performing the work or other activities (for example, it took extra effort) | 1 | 2 | 3 | 4 | 5 |
| | activities (for example, it took extra ellort) | | | | | |
| 12 | During the past 4 weeks, to what extent hinterfered with your normal social activitie | | | | | |
| 12 | During the <u>past 4 weeks</u> , to what extent he interfered with your normal social activities 1- Not at all | | | | | |
| 12 | During the <u>past 4 weeks</u> , to what extent he interfered with your normal social activities | | | | | |
| 12 | During the past 4 weeks, to what extent hinterfered with your normal social activities 1- Not at all 2- Slightly 3- Moderately 4- Quite a bit | | | | | |
| 12 | During the past 4 weeks, to what extent hinterfered with your normal social activities 1 Not at all 2- Slightly 3- Moderately | | | | | |



#### CASA-Q USER'S AGREEMENT

between Boehringer Ingelheim International GmbH, at Binger Str. 173, 55216 Ingelheim am Rhein, Germany (hereinafter "BOEHRINGER") and Hospital Canselor Tuanku Muhriz, Universiti Kebangsaan Malaysia, Jalan Yaacob Latiff, Bandar Tun Razak, 56000 Cheras, Kuala Lumpur, Malaysia (hereinafter "Licensee").

BOEHRINGER hereby grants permission to the Licensee to employ the Cough and Sputum Assessment Questionnaire (CASA-Q) in a study entitled "A Randomised, Open Label, Interventional Study Evaluating the Efficacy & Safety of Dry Powder Ivy Extract (Syrup Prospan) Vs NAC among COPD Patients". Licensee will be supported by Delfi Marketing Sdn Bhd, Level 6, Block A, Sky Park One City, Jalan USJ 25/1, 47650 Subang Jaya, Selangor, Malaysia to perform the study. Study results will be owned by Licensee.

BOEHRINGER will supply the Licensee with the CASA-Q in its original version (US English) and currently available translations, as listed below.

#### none

CASA-Q User Agreement

The instrument will be administered on paper. The Licensee acknowledges that new translations must be carried out by ICON/MAPI.

The use of the CASA-Q in the above-mentioned study to the following conditions:

| Th | e study is intended to be performed with 120 patients. |
|---|---|
| | For commercial studies the permission to use the CASA-Q is granted with a royalty fee of US\$ $5.00$ per patient. |
| | The Licensee will pay a royalty fee in the amount of US\$ 0.00 (nil USD) to BOEHRINGER for use of the CASA-Q in this study. Payment is due within 60 days upon signature of this Agreement by authorized representatives from both parties. |
| | Sponsors of new translations will be exonerated from the royalty fee. This means, the Licensee can use the existing translations in this study at no charge. |
| ☑ | The use of the CASA-Q in academic research or individual clinical practice is free of charge. |
| use | e CASA-Q is a copyrighted questionnaire owned by BOEHRINGER and must be<br>ad in its entirety. The Licensee, therefore, must not modify, abridge, translate, adapt<br>transform the CASA-Q in any manner or form without the prior written consent of |

July 8, 2023

BOEHRINGER. If such consent is given the copyright in such modifications, abridgments, translations, adaptations or transformations shall be vested exclusively in Boehringer Ingelheim International GmbH. The Licensee confirms that on each copy of the CASA-Q the copyright will be stated as "Copyright by Boehringer Ingelheim International GmbH 2008".

- The Licensee will not reproduce the CASA-Q except for the limited purpose of generating sufficient copies for the use in the study and shall in no event distribute copies of the CASA-Q to third parties by sale, rental, lease, lending, or any other means.
- The Licensee shall retain all rights to any data and/or results generated by the use of CASA-Q in the study.
- 4. The Licensee is free to publish any results of the study provided that Licensee does not publish any part of the CASA-Q and that all publications include the copyright clause as stated in Article 1.
- This Agreement holds for the above-mentioned study only. The use of the CASA-Q in any additional study of the Licensee will require a separate agreement.
- The license period dates from the Effective Date (date of last signature) to one (1) year after completion of the study.
- Place of venue for all disputes arising in connection with this Agreement is Frankfurt.
   This Agreement is governed by German Law.
- 8. This Agreement may be executed in two or more counterparts, each of which shall be deemed an original and all of which shall together be deemed to constitute one agreement. The parties agree that execution of this Agreement by industry standard electronic signature software and /or by exchanging PDF signatures shall have the same legal force and effect as the exchange of original signatures. If any proceeding arising under or relating to this Agreement, each party hereby waives any right to raise any defense or waiver based upon execution of this Agreement by means of such electronic signatures or maintenance of the executed agreement electronically

Signed and dated by: 11-Jul-2023 Boehringer Ingelheim International GmbH

i.V. i.

Dr. Karin Becker

Or. Karin Becker

Dr. Karin Becker

Dagmar Kaschinski

Signed and dated by: Hospital Canselor Tuanku Muhriz

Associate Prof Dr Mohamed Faisal Abdul Hamid

Consultant Pulmonologist Faculty of Medicine

Hospital Canselor Tuanku Muhriz Universiti Kebangsaan Malaysia

11 July 2023

2

CASA-Q User Agreement

July 8, 2023

#### **Section 14: References**

- 1. World Health Organization. Chronic obstructive pulmonary disease (COPD). www.who.int/news-room/fact-sheets/detail/chronic-obstructive-pulmonary-disease-(copd) Date last accessed: 27 May 2022. Date last updated: 20 May 2022
- 2. BD 2017 DALYs and HALE Collaborators. Global, regional, and national disability-adjusted life-years (DALYs) for 359 diseases and injuries and healthy life expectancy (HALE) for 195 countries and territories, 1990–2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet 2018; 392: 1859–1922. doi:10.1016/S0140-6736(18)32335-3
- 3. Seemungal TA, Hurst JR, Wedzicha JA. Exacerbation rate, health status and mortality in COPD--a review of potential interventions. Int J Chron Obstruct Pulmon Dis 2009; 4: 203–223. doi:10.2147/copd.s3385
- 4. Donaldson GC, Wedzicha JA. COPD exacerbations. 1: Epidemiology. Thorax 2006; 61: 164–168. doi:10.1136/thx.2005.041806
- 5. Donaldson GC, Law M, Kowlessar B, et al. Impact of prolonged exacerbation recovery in chronic obstructive pulmonary disease. Am J Respir Crit Care Med 2015; 192: 943–950. doi:10.1164/rccm.201412-2269OC
- 6. Curran DR, Cohn L. Advances in mucous cell metaplasia: a plug for mucus as a therapeutic focus in chronic airway disease. Am J Respir Cell Mol Biol 2010; 42: 268–275. doi:10.1165/rcmb.2009-0151TR
- 7. Poole P, Sathananthan K, Fortescue R. Mucolytic agents versus placebo for chronic bronchitis or chronic obstructive pulmonary disease. Cochrane Database Syst Rev 2019; 5: CD001287. doi:10.1002/14651858.CD001287.pub6
- 8. Rogers DF. Mucoactive drugs for asthma and COPD: any place in therapy? Expert Opin Investig Drugs 2002; 11: 15–35.
- 9. Du Y, Wolf IK, Zhuang W, Bodemann S, Knoss W, Knopf H. Use of herbal medicinal products among children and adolescents in Germany. BMC Complement Altern Med. 2014;14(218):218. doi: 10.1186/1472-6882-14-218.
- 10. European Medicines Agency Committee on Herbal Medicinal Products (HMPC) (2018) Assessment report on Hedera helix L., folium
- 11. R. Balsamo, L. Lanata, C. G. Egan. Mucoactive drugs. European Respiratory Review 2010 19: 127-133; DOI: 10.1183/09059180.00003510

- 12. Linden M, Wieslander E, Eklund A, *et al.* Effects of oral *N*-acetylcysteine on cell content and macrophage function in bronchoalveolar lavage from healthy smokers. *Eur Respir J* 1988; 1: 645–650.
- 13. Niederman MS, Rafferty TD, Sasaki CT, *et al.* Comparison of bacterial adherence to ciliated and squamous epithelial cells obtained from the human respiratory tract. *Am Rev Respir Dis* 1983; 127: 85–90.
- 14. Efthymia Papadopoulou, Jan Hansel, Zsofia Lazar, Konstantinos Kostikas, Stavro s Tryfon, Jørgen Vestbo, Alexander G. Mathioudakis, European Respiratory Review 2023 32: 220141; DOI: 10.1183/16000617.0141-2022
- 15. Mario Cazzola 1, Paola Rogliani 1, Luigino Calzetta 1, Nicola A Hanania 2, Maria Gabriella Matera 3 COPD. 2017 Oct;14(5):552-563. doi: 10.1080/15412555.2017.1347918. Epub 2017 Jul 28.
- 16. Völp, A., Schmitz, J., Bulitta, M. *et al.* Ivy leaves extract EA 575 in the treatment of cough during acute respiratory tract infections: meta-analysis of double-blind, randomized, placebo-controlled trials. *Sci Rep* 12, 20041 (2022). <a href="https://doi.org/10.1038/s41598-022-24393-1">https://doi.org/10.1038/s41598-022-24393-1</a>
- 17. Karel Kostev, Andreas Völp, Fanny Ludwig, Christoph Strehl & Georg Seifert (2022) Association between ivy leaves dry extract EA 575 prescriptions and antibiotic use, sick leave duration, and repeated infections in adult patients, Postgraduate Medicine, 134:3, 333 340, DOI: 10.1080/00325481.2022.2015220
- 18. Rogliani P, Matera MG, Page C, Puxeddu E, Cazzola M, Calzetta L. Efficacy and safety profile of mucolytic/antioxidant agents in chronic obstructive pulmonary disease: a comparative analysis across erdosteine, carbocysteine, and Nacetylcysteine. Respir Res 2019; 20(1): 104
- 19. Cohen, J. (1998) Statistical Power Analysis for the Behavioural Sciences. Lawrence Erlbaum Associates, Hillsdale.
- 20. Kuzmenko, N., Iaremenko, O., Dobrianskiy, D., Ilnytskyi, R., and Gumeniuk, G. (2020). The efficacy and safety of inhaled acetylcysteine in comparison with oral acetylcysteine in chronic obstructive pulmonary disease: A randomized single-center study. Polish Annals of Medicine, 27(2), pp.108-114. https://doi.org/10.29089/2020.20.00112
- 21. Dhand, N. K., & Khatkar, M. S. (2014). Statulator: An online statistical calculator. Sample Size Calculator for Comparing Two Paired Means. Accessed 6 June 2023 at http://statulator.com/SampleSize/ss2PM.html